CLINICAL TRIAL: NCT02135614
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Multi-Center Study Evaluating Antiviral Effects, Pharmacokinetics, Safety, and Tolerability of GS-5806 in Hospitalized Adults With Respiratory Syncytial Virus (RSV) Infection
Brief Title: Efficacy, Pharmacokinetics, and Safety of Presatovir in Hospitalized Adults With Respiratory Syncytial Virus (RSV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-218-1227; 2014-002137-58 (EudraCT Number)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Presatovir (Experimental): Participants will receive a single dose of presatovir.
  Interventions: Drug: Presatovir
- Presatovir placebo (Placebo Comparator): Participants will receive a single dose of presatovir placebo.
  Interventions: Drug: Presatovir placebo

INTERVENTIONS:
Drug: Presatovir — Presatovir 200 mg (4 x 50 mg tablets) administered orally
  Other Names: GS-5806
  Arms: Presatovir
Drug: Presatovir placebo — Presatovir placebo tablets administered orally
  Arms: Presatovir placebo

SUMMARY:
The primary objective of this study is to evaluate the effects of presatovir on respiratory syncytial virus (RSV) viral load in RSV-positive adults who have been hospitalized with acute respiratory infectious symptoms.

Participants will receive 1 dose of presatovir on Day 1 and followed for 27 days postdose. Nasal swabs will be collected at each study visit (excluding Day 28) and assayed for change in viral load as the primary endpoint.

ELIGIBILITY:
Key Inclusion Criteria:

* Current inpatient
* New onset of acute respiratory infectious symptoms, or acute worsening of chronic symptoms related to ongoing respiratory disease for ≤ 5 days prior to screening:

  * Upper respiratory tract symptoms: nasal congestion, runny nose, sore throat, or earache
  * Lower respiratory tract symptoms: cough, sputum production, wheezing, dyspnea, or chest tightness
* Documented to be RSV-positive at the current admission within 72 hours of screening, or as evaluated at screening

Key Exclusion Criteria:

* Related to concomitant or previous medication use:

  * Use of oral prednisone or other corticosteroid equivalent to:

    * > 20 mg/day for > 14 days prior to screening is not permitted.
    * > 20 mg/day for ≤ 14 days, including corticosteroids received during current hospitalization (ie, bolus doses), is permitted.
    * ≤ 20 mg/day, regardless of duration, is permitted.
  * Individuals taking a moderate or strong cytochrome P450 enzyme (CYP) inducer including but not limited to rifampin, St John's Wort, carbamazepine, phenytoin, efavirenz, bosentan, etracirine, modafinil, and nafcillin within 2 weeks prior to the first dose of study drug
* Related to medical history:

  * Pregnant, breastfeeding, or lactating females
  * Individuals requiring > 50% supplemental oxygen (while the individual is awake) at screening
  * Individuals with a Clinical Frailty Scale (CFS) > 7 at Baseline
  * Known significant abnormality altering the anatomy of the nose or nasopharynx that in, the opinion of the investigator, will preclude obtaining adequate nasal swab sampling in either nasal passage
  * Waiting for or recently (within the past 12 months) received a bone marrow, stem cell, or solid organ transplant, or who have received radiation or chemotherapy within 12 months prior to Screening
  * Individuals with HIV/AIDS and a known CD4 count < 200 cells/uL
  * History of severe dementia or Alzheimer's disease
  * History of drug and/or alcohol abuse that, in the opinion of the investigator, may prevent adherence to study activities
* Related to medical condition at screening:

  * Influenza-positive as determined by local diagnostic test
  * Known Middle East Respiratory Syndrome coronavirus (MERS-CoV) infection or known coinfection with other coronavirus
  * Use of mechanical ventilation during the current admission, not including noninvasive ventilation
  * Clinically significant bacteremia or fungemia that has not been adequately treated prior to Screening, as determined by the investigator
  * Inadequate treatment of confirmed bacterial, fungal, or non-RSV pneumonia, as determined by the investigator
  * Excessive nausea/vomiting at admission, as determined by the investigator, that precludes administration of an orally administered study drug
* Related to allergies:

  * Known allergy to components of the study drug (microcrystalline cellulose, mannitol, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol and talc)
  * Documented history of acute (anaphylaxis) or delayed (Stevens-Johnson syndrome or epidermal necrolysis) allergy to sulfa drugs

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (43):
- United States (9):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont, Royal Oak, Michigan
  - New York Presbyterian Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Vanderbilt Medical Group and Clinic, Nashville, Tennessee
  - University of Washington, Seattle, Washington
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Australia (6):
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Monash Medical Center, Clayton, Victoria
  - Frankston Hospital, Frankston, Victoria
- Universite Liebre de Bruxelles - Hopital Erasme, Anderlecht, Belgium
- France (6):
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - CHRU Brest - Hospital Cavale Blanche, Brest
  - Hopital d'Instructions des Armees Percy, Clamart
  - Hopital Louis Mourier, Colombes
  - Hopital Saint Louis - Service de Pneumologie, Paris
  - Hopital Tenon, Paris
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Edith Wolfson Medical Center, Holon
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Western Galilee Hospital-Nahariya, Nahariya
  - The Nazareth Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
- Gelre Ziekenhuizen, Zutphen, Netherlands
- New Zealand (3):
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Middlemore Hospital, Auckland
  - Waikato Hospital, Hamilton
- Centrum Badan Klinicznych, Wroclaw, Poland
- South Korea (4):
  - Soon Chun Hyang University Hospital, Bucheon-si
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- United Kingdom (2):
  - Southampton University Hospitals NHS Trust, Southampton
  - Princess Royal Hospital, Telford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, Asia, New Zealand, and the United States. The first participant was screened on 09 June 2014. The last study visit occurred on 12 April 2017.
Pre-assignment Details: 833 participants were screened.
Groups:
- Presatovir: Single dose of presatovir 200 mg (4 x 50 mg tablets)
- Placebo: Single dose of placebo tablets
Period: Overall Study
Arm/Group | Presatovir | Placebo
Started | 94 | 95
Completed | 86 | 90
Not Completed | 8 | 5
Not completed — Randomized but Not Treated | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Investigator's Discretion | 0 | 1
Not completed — Withdrew Consent | 2 | 2
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Presatovir | Placebo | Total
Number analyzed (Participants) | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (14.24) | 65.9 (13.87) | 67.6 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 42 | 42 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 11 | 17
  Black or African American | 5 | 7 | 12
  Native Hawaiian or Pacific Islander | 0 | 2 | 2
  White | 72 | 69 | 141
  Other | 2 | 2 | 4
  Not Permitted | 7 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 85 | 91 | 176
  Not Permitted | 7 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 9 | 9 | 18
  Netherlands | 0 | 2 | 2
  South Korea | 5 | 11 | 16
  Belgium | 0 | 1 | 1
  United States | 15 | 14 | 29
  Poland | 1 | 5 | 6
  Italy | 1 | 0 | 1
  United Kingdom | 1 | 4 | 5
  Israel | 32 | 26 | 58
  Australia | 10 | 5 | 15
  France | 18 | 17 | 35
Stratification Factor: Disease Status [Count of Participants; unit: Participants]
  Asthma | 22 | 22 | 44
  Chronic Obstructive Pulmonary Disease | 27 | 30 | 57
  No Chronic Airways or Lung Disease | 31 | 31 | 62
  Other Chronic Airways or Lung Disease | 12 | 11 | 23
Nasal Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 5.58 (2.104) | 5.07 (2.528) | 5.32 (2.337)
Flu-PRO score [Mean (Standard Deviation); unit: units on a scale] — Flu-PRO Score was calculated as the mean of 38 individual scores. Individual scores ranged from 0 (no symptoms) to 4 (worst symptoms).
  units on a scale | 1.11 (0.553) | 1.04 (0.566) | 1.07 (0.559)
Duration of Hospitalization Prior to First Dose [Mean (Standard Deviation); unit: days] — Duration of hospitalization prior to the first dose date of study drug was calculated as (the first dose date - the admission date of hospitalization).
  days | 2.9 (3.14) | 3.2 (7.13) | 3.0 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change in Respiratory Syncytial Viral (RSV) Load From Baseline to Day 5
Description: The time-weighted average change, often referred to as the DAVG, provides the average viral burden change from baseline. The mean values presented were calculated using the ANCOVA model and are adjusted for baseline value and stratification factor.
Time Frame: Baseline to Day 5
Population: Evaluable Analysis Set: all randomized participants who received at least 1 dose of study medication, had an RSV viral load greater than lower limit of quantification (LLOQ) of the RT-qPCR assay in the Day 1 nasal-swab sample, and had a minimum of 3 quantifiable samples (including baseline) within a 5 day period.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 80 | 74
log10 copies/mL | -0.77 (0.113) | -0.89 (0.118)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.46, ANCOVA — P-value was calculated from the ANCOVA model including baseline values, Clinical Frailty Scale (CFS) score, and stratification factor as covariates; Treatment difference = 0.12, 95% CI 2-sided [-0.20 to 0.43]

2. Secondary Outcome: Time-weighted Average Change in the Flu-PRO Score From Baseline to Day 5
Description: The Flu-PRO is a patient-reported outcome questionnaire utilized as a standardized method for evaluating symptoms of influenza. Flu-PRO Score was calculated as the mean of 38 individual scores. Individual scores ranged from 0 (no symptoms) to 4 (worst symptoms). The mean values presented were calculated using the ANCOVA model and are adjusted for baseline value and stratification factor.
Time Frame: Baseline to Day 5
Population: Participants in the Evaluable Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 79 | 74
units on a scale | -0.27 (0.029) | -0.35 (0.030)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.046, ANCOVA — P-value was calculated from the ANCOVA model including the baseline value, CFS score and stratification factor as covariates; Treatment difference = 0.08, 95% CI 2-sided [0.00 to 0.16]

3. Secondary Outcome: Number of Hospitalization-Free Days Following Presatovir Administration
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 80 | 74
days | 25 [20 to 27] | 25 [20 to 27]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.39, Negative Binomial Model — P-value was calculated from the negative binomial model with the stratification factor as covariate

4. Secondary Outcome: Rate of Unplanned Medical Encounters
Description: The adjusted rate of unplanned medical encounters (clinic visits, emergency room visits, urgent care visits, and rehospitalizations) related to a respiratory illness after initial hospital discharge through Day 28 will be assessed. Event rate was calculated as the total number of unplanned medical encounters divided by the total number of participants. The mean values presented were adjusted for stratification factor.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: encounters per participant
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 80 | 74
encounters per participant | 0.226 [0.133 to 0.384] | 0.066 [0.029 to 0.150]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.004, Negative Binomial Model — P-value from the negative binomial model comparing the rate ratio between treatment groups, adjusted for the stratification factor

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety Analysis Set: all participants who received 1 dose of study drug.
Arm/Group | Presatovir | Placebo
All-Cause Mortality (participants affected / at risk) | 2/92 | 0/94
Serious Adverse Events (participants affected / at risk) | 8/92 | 13/94
Other Adverse Events (participants affected / at risk) | 34/92 | 31/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=92) | Placebo (N=94)
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=92) | Placebo (N=94)
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 4 | 9
Vomiting (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 5 | 1
Alanine aminotransferase increased (Investigations) | 5 | 2
Headache (Nervous system disorders) | 8 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (6):
  • Study Protocol: Original (2013-11-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/Prot_006.pdf
  • Study Protocol: Amendment 1 (2014-03-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/Prot_007.pdf
  • Study Protocol: Amendment 2 (2014-08-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/Prot_008.pdf
  • Study Protocol: Amendment 3 (2014-08-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/Prot_009.pdf
  • Study Protocol: Amendment 4 (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/Prot_010.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02135614/SAP_011.pdf